CLINICAL TRIAL: NCT06617507
Title: The Effect of Selective Dorsal Rhizotomy Surgery on Walking in Children With Ambulatory Cerebral Palsy in Turkey
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Gizem Gurzoglu, Pediatric Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: GGurzoglu2
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy Spastic Diplegia; Gait, Spastic
Keywords: Cerebral Palsy; Gait; Selective Dorsal Rhizotomy; Ambulation
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with diparetic cerebral palsy: 20 ambulatory diparetic CP cases were included. The Modified Ashworth Scale (MAS), The Gillette Functional Assessment Questionnaire (FAQ) and The Edinburgh Visual Gait Score (EVGS) were applied to the participants.
  Interventions: Other: Group 1

INTERVENTIONS:
Other: Group 1 — The Modified Ashworth Scale (MAS), The Gillette Functional Assessment Questionnaire (FAQ) and The Edinburgh Visual Gait Score (EVGS) were applied to the participants.

SUMMARY:
Cerebral Palsy (CP) is a motor disorder that develops during fetal brain development or due to non-progressive damage to the developing infant brain. These movement and posture disorders are classified as Spastic Type, Dyskinetic Type, Ataxic Type and Mixed Type (Rosenbaum, 2007). Spastic type CP accounts for 20% of all CP cases. Spastic type CP is divided into three groups: diparetic (38%), hemiparetic (39%) and quadriparetic (23%) (Novak et al., 2014).

Lower extremity involvement is more common in diparetic cerebral palsy (DCP) (Donker et al., 2008). 98% of DCP cases vary between GMFS levels I and III. Walking rates are between 86-91% (Novak et al., 2014). Children with DCP can usually walk until the age of 4 (Cottalorda, 1998). However, these walks are often; Due to spasticity, muscle weakness, involuntary co-contraction, deficiencies in selective motor control, balance problems, structural changes of soft tissue and compensatory mechanisms (Manca, 2014), it can lead to musculoskeletal system problems and gait pathologies. Although the cerebral lesion that causes is static, children with spastic diplegia increase in height with age, and they may lose their ability to walk because bone length cannot be accompanied by muscle length at the same rate (Miller, 2020).

Selective Dorsal Rhizotomy (SDR) surgery is an effective method for spasticity management in children with spastic DCP (Novak et al., 2014). The positive effect of SDR on function and mobility has been proven (Novak et al., 2020).

It has been stated that SDR surgery applied to carefully selected candidates may be beneficial on gait quality in individuals with ambulatory CP (Chen, 2019). SDR surgery has been found to improve walking as a result of information collected from patients through a survey (Park, 2021). The aim of our study is to reveal the effect of SDR surgery performed in Turkey on gait function in children with CP using evaluation scales.

DETAILED DESCRIPTION:
It's an observational study. Purpose of the study: The aim of our study is to reveal the effect of SDR surgery performed in Turkey on gait function in children with CP using evaluation scales.

A total of 20 ambulatory diparetic CP cases, aged between 0-17, who were deemed suitable for SDR surgery and operated on, were included in the study.

* What is the effect of SDR surgery performed in Turkey on gait function in children with CP?
* How did the muscle tone of the participants change after the SDR operation?

The Modified Ashworth Scale (MAS), The Gillette Functional Assessment Questionnaire (FAQ) and The Edinburgh Visual Gait Score (EVGS) were applied to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 0-17
* Being diagnosed with Diparetic CP, one of the types of Cerebral Palsy

Exclusion Criteria:

* Having any history of orthopedic surgery on the musculoskeletal system
* Having Botulinum Toxin injection in the last 6 months
* Using of Baclofen Pump

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 20 ambulatory diparetic CP cases, aged between 0-17, who were deemed suitable for SDR surgery and operated on, were included in the study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The Modified Ashworth Scale (MAS) | baseline
  It is a 6-point scale used to describe the muscle's resistance to passive movement and the ease with which the joint can be moved within the available range. It is frequently used in clinical settings. Its evaluation and interpretation are quite practical. Within the scope of the study, lower extremity muscles were evaluated with MAS.
The Gillette Functional Assessment Questionnaire (FAQ) | baseline
  It is a measurement tool used to evaluate walking ability and functional mobility in children. This questionnaire was developed specifically to evaluate the walking functions of children with CP and other neuromuscular disorders. Developed at Gillette Children's Hospital, this survey aims to rate children's walking abilities in different environments. Scores children's walking skills between 1-10.
The Edinburgh Visual Gait Score (EVGS) | baseline
  EVGS is a valid and reliable gait analysis method used in gait evaluation in children with CP. It is a practically used gait analysis that supports observational gait analysis, especially in children with CP with mild involvement and distal deformities. In EVGS, evaluation is made by video recording method. It consists of 17 parameters and evaluates gait in frontal, sagittal and transverse planes. In each lower extremity, 6 anatomical regions, namely trunk, pelvis, hip, knee, ankle and foot, are evaluated separately during the stance and swing phases of gait.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Gürzoğlu, Study Director — Acıbadem Atunizade Hospital
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Altunizade, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.